CLINICAL TRIAL: NCT06585072
Title: Prospective Cohort Study on Endo-Exdo Secretory Function Alterations and All-round Outcomes After Pancreatic Cancer
Brief Title: Pancreatic Cancer and Diabetes Mellitus
Status: Recruiting | Type: Observational
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Tuo Li, MD, Deputy Director, Shanghai Changzheng Hospital
Other Study IDs: NMU-3CDM-2B
Record Dates: First submitted 2024-09-02; First posted 2024-09-05 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Cancer; Surgery; Diabetes Mellitus
Keywords: Pancreatic Cancer; Surgery; Diabetes Mellitus; Risk factor
MeSH Terms: conditions — Pancreatic Neoplasms; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples will be collected at every visit
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: All enrolled subjects completed dynamic blood glucose monitoring to obtain continuous peripheral blood glucose data. — All enrolled subjects completed dynamic blood glucose monitoring to obtain continuous peripheral blood glucose data.

SUMMARY:
The goal of this observational study is to learn about post-surgery of pancreatic cancer diabetes mellitus.The main questions it aims to answer are:

1. Are the incident rates of glucose metabolic disorders (pre-diabetes and diabetes mellitus) after pancreatic cancer of different etiologies the same?
2. Are alterations in endocrine and exdocrine secretory function in patients with pancreatic surgery associated with all-round outcomes? All patients with pancreatic surgery have been given the standardized treatment for the condition.

The reasearchers will summarize the incident rates of glucose metabolic disorders (pre-diabetes and diabetes mellitus) during different surgical procedures to explore the association between alternations in endocrine and exdocrine secrectory function and all-round outcomes.

DETAILED DESCRIPTION:
Investigators will prospectively collect data from patients with pancreatic cancer after surgery in participant centers.

ELIGIBILITY:
Inclusion Criteria:

1. male or female Chinese subjects; 2. Age ≥ 18 years; 3. patients with pancreatic cancer who are proposed to undergo pancreatectomy by pancreaticobiliary surgery at our hospital; 4. those who voluntarily completed the Pancreatobiliary Surgery Cohort Study and signed the informed consent; 5. those who have completed and banked serum and pathological specimens at our hospital.

-

Exclusion Criteria:

1. those with a previous history of comorbid diabetes mellitus or pre-diabetes mellitus, or preoperative HbA1C ≥ 6.0% or fasting blood glucose ≥ 6.1 mmol/l; 2. those with positive islet-associated antibodies 3. those with the presence of medications, endocrine disease exposures that can lead to a risk of secondary diabetes; 4. pregnant or nursing women; 5. Cognitive impairment or other reasons for failing to sign the informed consent form.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pancreatic cancer after pancreatic surgery
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who developed glucose metabolic disorders(pre-diabetes and diabetes mellitus) | From enrollment to five years after the end of the surgery
  The diagnosis of glucose disorders should be made applying criteria of the American Diabetes Association.

SECONDARY OUTCOMES:
Overall Survival | From enrollment to five years after the end of the surgery
Disease-Free Survival | From enrollment to five years after the end of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: tuo Li, Prof., Study Director — Shanghai Changzheng Hospital
Locations (1):
- Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No